CLINICAL TRIAL: NCT02279095
Title: A Phase 2, Open-Label Extension, Efficacy and Safety Study of a Retinoic Acid Receptor Gamma (RARγ) Specific Agonist (Palovarotene) in the Treatment of Preosseous Flare-ups in Subjects With Fibrodysplasia Ossificans Progressiva (FOP)
Brief Title: An Open-Label Extension Study of Palovarotene Treatment in Fibrodysplasia Ossificans Progressiva (FOP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVO-1A-202; 2014-002496-28 (EudraCT Number); NCT02979769 (obsolete NCT alias)
Record Dates: First submitted 2014-10-26; First posted 2014-10-30 (Estimated); Results first posted 2024-05-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Fibrodysplasia Ossificans Progressiva
Keywords: Open-label extension study; Clinical trial Phase 2; Efficacy and safety; Heterotopic ossification; Fibrodysplasia Ossificans Progressiva; Flare-up; Palovarotene; Retinoic acid receptor agonist; Retinoic acid receptor gamma agonist; Clementia; Myositis Ossificans Progressiva; Munchmeyer's Disease; FOP; Ipsen
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Palovarotene dose level 1 (completed) (Experimental): Participants received 10 mg palovarotene for 14 days, followed by 5 mg palovarotene for 28 days (or weight-based equivalent) for eligible flare-ups (Part A).
  Interventions: Drug: Palovarotene dose level 1
- Palovarotene dose level 2 (Experimental): Participants with at least 90% skeletal maturity received 5 mg palovarotene for up to 24 months and 20 mg palovarotene for 28 days, followed by 10 mg for 56 days for eligible flare-ups (Part B).
  Interventions: Drug: Palovarotene dose level 2
- Palovarotene dose level 3 (Experimental): Participants with less than 90% skeletal maturity received weight-adjusted doses of 20 mg palovarotene for 28 days, followed by 10 mg for 56 days for eligible flare-ups (Part B).
  Interventions: Drug: Palovarotene dose level 3
- Palovarotene dose level 4 (Experimental): All participants will receive 5 mg palovarotene for up to 48 months and 20 mg palovarotene for 28 days, followed by 10 mg for 56 days for eligible flare-ups (Part C). Skeletally immature participants will receive weight-adjusted doses.
  Interventions: Drug: Palovarotene dose level 4

INTERVENTIONS:
Drug: Palovarotene dose level 1 — Palovarotene was taken orally once daily at approximately the same time each day.
  Arms: Palovarotene dose level 1 (completed)
Drug: Palovarotene dose level 2 — Palovarotene will be taken orally once daily at approximately the same time each day.
  Arms: Palovarotene dose level 2
Drug: Palovarotene dose level 3 — Palovarotene will be taken orally once daily at approximately the same time each day.
  Arms: Palovarotene dose level 3
Drug: Palovarotene dose level 4 — Palovarotene will be taken orally once daily at approximately the same time each day.
  Arms: Palovarotene dose level 4

SUMMARY:
Fibrodysplasia Ossificans Progressiva (FOP) is a rare, severely disabling disease characterized by heterotopic ossification (HO), i.e., abnormal bone formation, often associated with painful, recurrent episodes of soft tissue swelling (flare-ups). Lesions begin in early childhood and lead to progressive ankyloses of major joints with resultant loss of movement.

In this study, the ability of different palovarotene dosing regimens to prevent the formation of new HO will be evaluated in adult and pediatric participants with FOP.

DETAILED DESCRIPTION:
The main objective of this Phase 2, multicenter, open-label study is to evaluate the safety and efficacy of different palovarotene dosing regimens in participants with FOP. Efficacy will be assessed based on the ability of palovarotene to prevent the formation of new heterotopic ossification (HO) as assessed by low-dose whole body computed tomography (WBCT) scan, excluding head.

The study was divided into four parts: Part A (completed on July 2017), Part B (completed on October 2018), Part C (completed) and Part D (completed). Each part was associated with revised palovarotene treatment regimens.

In Part A, all pediatric and adult participants who successfully completed Study PVO-1A-201 were enrolled and followed for up to 36 months. Participants who had an eligible flare-up received 10 mg palovarotene daily for 14 days, followed by 5 mg palovarotene daily for 28 days (or weight-based equivalent).

In Part B, participants who successfully completed Study PVO-1A-201 (including any participant who participated in Part A of Study PVO-1A-202) as well as up to 20 new adult participants were followed for up to 24 months. The Adult Cohort included all participants with at least 90% skeletal maturity, regardless of age. The Pediatric Cohort included all participants with less than 90% skeletal maturity. Any Pediatric Cohort participant who achieved ≥90% skeletal maturity during Part B was considered for enrollment into the Adult Cohort at the discretion of the Investigator. Part B added a 5 mg palovarotene daily chronic treatment regimen administered between flare-ups for participants in the Adult Cohort for up to 24 months. Part B also increased the flare-up dosing to 20 mg palovarotene daily for 28 days, followed by 10 mg palovarotene daily for 56 days (or weight-adjusted equivalents in the Pediatric Cohort). Treatment could be extended if the flare-up was still ongoing.

In Part C, participants from Part B are being followed for up to an additional 48 months. There will be no new participants in Part C. All eligible participants, including skeletally immature participants, are receiving 5 mg palovarotene daily chronic treatment regimen (weight-adjusted doses for skeletally immature participants).

In Part D, annual post last dose of study treatment assessments for up to 2 years will be obtained in participants who were skeletally immature at the time of study treatment discontinuation in order to obtain longer-term safety data. No new participants will be enrolled into Part D.

Part C plus Part D duration will not exceed 48 months.

All participants will undergo all study procedures as specified in the respective schedule of assessments and for as long as they are not 100% skeletally mature.

ELIGIBILITY:
Inclusion Criteria:

* Completion of Study PVO-1A-202/Part B.
* Written, signed, and dated informed consent and, for participants who are minors, age-appropriate participant assent (performed according to local regulations).
* Accessible for treatment with palovarotene and follow-up (able and willing to travel to a site for the initial and all follow-up clinic visits).
* Able to undergo low-dose, WBCT scan, excluding head.
* Females of child-bearing potential must have a negative blood or urine pregnancy test (with sensitivity of at least 50 mIU/mL) prior to administration of palovarotene.
* Male and FOCBP participants must agree to remain abstinent from heterosexual sex during treatment and for 1 month after treatment or, if sexually active, to use two effective methods of birth control during and for 1 month after treatment. Additionally, sexually active females of childbearing potential (FOCBP) participants must already be using two effective methods of birth control 1 month before treatment is to start. Specific risk of the use of retinoids during pregnancy, and the agreement to remain abstinent or use two effective methods of birth control will be clearly defined in the informed consent and the participant or legally authorized representatives.

Exclusion Criteria:

* Any reason that, in the opinion of the Investigator, would lead to the inability of the participant and/or family to comply with the protocol.
* Amylase or lipase >2x above the upper limit of normal or with a history of pancreatitis.
* Elevated aspartate aminotransferase or alanine aminotransferase >2.5x the upper limit of normal.
* Fasting triglycerides >400 mg/dL with or without therapy.
* Currently using vitamin A or beta carotene, multivitamins containing vitamin A or beta carotene, herbal preparations containing vitamin A or beta carotene, or fish oil, and unable or unwilling to discontinue use of these products during palovarotene treatment.
* Participants experiencing suicidal ideation (type 4 or 5) or any suicidal behavior within the past month as defined by the Columbia Suicide Severity Rating Scale (C-SSRS).

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- United States (3):
  - University of California San Francisco, Division of Endocrinology and Metabolism, San Francisco, California
  - Mayo Clinic, Department of Medicine, Rochester, Minnesota
  - University of Pennsylvania, Center for FOP & Related Bone Disorders, Philadelphia, Pennsylvania
- Hospital Italiano de Buenos Aires, Department of Pediatrics, Buenos Aires, Argentina
- Australia (2):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Queensland University of Technology (QUT) Institute of Health and Biomedical Innovation (IHBI), Woolloongabba, Queensland
- Hôpital Necker-Enfants Malades, Department of Genetics, Paris, France
- The Royal National Orthopaedic Hospital, Brockley Hill, Stanmore, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shimono K, Tung WE, Macolino C, Chi AH, Didizian JH, Mundy C, Chandraratna RA, Mishina Y, Enomoto-Iwamoto M, Pacifici M, Iwamoto M. Potent inhibition of heterotopic ossification by nuclear retinoic acid receptor-gamma agonists. Nat Med. 2011 Apr;17(4):454-60. doi: 10.1038/nm.2334. Epub 2011 Apr 3. PMID 21460849
- [Derived] Pignolo RJ, Al Mukaddam M, Baujat G, Brown MA, De Cunto C, Hsiao EC, Keen R, Le Quan Sang KH, Grogan DR, Marino R, Strahs AR, Kaplan FS. Study methodology and insights from the palovarotene clinical development program in fibrodysplasia ossificans progressiva. BMC Med Res Methodol. 2023 Nov 13;23(1):269. doi: 10.1186/s12874-023-02080-7. PMID 37957586
- [Derived] Pignolo RJ, Kimel M, Whalen J, Kawata AK, Artyomenko A, Kaplan FS. The Fibrodysplasia Ossificans Progressiva Physical Function Questionnaire (FOP-PFQ): A patient-reported, disease-specific measure. Bone. 2023 Mar;168:116642. doi: 10.1016/j.bone.2022.116642. Epub 2022 Dec 13. PMID 36526263
- See also: Website for the International FOP Association — http://ifopa.org
- See also: Website for the French FOP Association — http://fopfrance.fr
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2024/02/14114118/Study-PVO-1A-202-Palovarotene-in-FOP-lay-summary.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2, open-label extension of study PVO-1A-201 was conducted in participants with FOP at 8 investigational sites in 5 countries. Participants enrolled in France were followed under a country-specific study PVO-1A-204 (as Part B of the study) as requested by French regulatory authorities. Overall, 58 participants were enrolled in this study.
Pre-assignment Details: Study divided into 4 parts: Part A (participants who completed PVO-1A-201 study were enrolled and followed for 3 years), Part B (participants from Part A and 18 new adult participants were followed for 2 years), Part C (participants from Part B were followed for 2 years) and Part D (treatment discontinued participants were followed for 2 years).
Groups:
- All Participants: Participants who completed PVO-1A-201 study were followed for up to 36 months in Part A. Eligible participants with a flare-up received palovarotene 10 milligram (mg) capsule orally daily for 2 weeks followed by 5 mg daily for 4 weeks during the flare-up component of Part A.
  In Part B, eligible participants from Part A and participants from the new Adult Cohort received chronic treatment with palovarotene 5 mg daily for up to 24 months. Participants with flare-ups received palovarotene 20 mg daily for 4 weeks followed by 10 mg daily for 8 weeks.
  In Part C, eligible participants received chronic treatment of palovarotene 5mg daily for up to 36 months. Participants with flare-ups received palovarotene 20 mg daily for 4 weeks followed by 10 mg daily for 8 weeks. For skeletal immature participants, the exposure-equivalent dose was determined based on weight.
  In Part D, no study drug was administered. Participants in Part C/D were followed for up to an additional 48 months.
Period: Overall Study
Arm/Group | All Participants
Started | 58
Entered Part A | 40
Completed Part A | 13
Entered Part B (New Adult Cohort into Part B) | 54
Completed Part B | 16
Entered Part C | 48
Completed Part C | 29
Entered Part D | 2
Completed | 39
Not Completed | 19
Not completed — Non-Compliance | 1
Not completed — Withdrawal by Subject | 8
Not completed — Adverse Event | 2
Not completed — Other | 7
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The Enrolled Population included all participants enrolled in the study.
Groups:
- All Participants: Participants who completed PVO-1A-201 study were followed for up to 36 months in Part A. Eligible participants with a flare-up received palovarotene 10 mg capsule orally daily for 2 weeks followed by 5 mg daily for 4 weeks during the flare-up component of Part A.
  In Part B, eligible participants from Part A and participants from the new Adult Cohort received chronic treatment with palovarotene 5 mg daily for up to 24 months. Participants with flare-ups received palovarotene 20 mg daily for 4 weeks followed by 10 mg daily for 8 weeks.
  In Part C, eligible participants received chronic treatment of palovarotene 5 mg daily for up to 36 months. Participants with flare-ups received palovarotene 20mg daily for 4 weeks followed by 10 mg daily for 8 weeks. For skeletal immature participants, the exposure-equivalent dose was determined based on weight.
  In Part D, no study drug was administered. Participants in Part C/D were followed for up to an additional 48 months.
Arm/Group | All Participants
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.0 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Parts A and B: Percentage of Flare-ups With No New Heterotopic Ossification (HO) at Week 12
Description: A responder was defined as a participant with no or minimal new HO at original flare-up site compared with baseline (pre-dose data from PVO-1A-201 study). Minimal new HO was defined as new HO with an HO score <=3 in both the anterior/posterior (AP) and lateral projections (or if 1 view is noninterpretable or non-evaluable, then remaining evaluable view was used). The HO score ranged from 0 to 6 where, 0 = no HO and 6 = single contiguous HO with longest dimension >2 diameters of reference normotopic bone in any projection. Highest HO score from 2 projections was used.
Time Frame: Baseline and Week 12
Population: Part A: Efficacy population included all participants in the treated population who had an evaluable Week 6 or Week 12 image [computed tomography (CT) scan or plain radiograph].
  Part B: Flare-up population included all participants in the treated population who took at least 1 dose of palovarotene during flare-up based treatment in Part B. Only participants with flare-ups at baseline and Week 12 are reported.
Measure: Number; unit: percentage of flare-ups
Units Other Than Participants: Flare-ups
Groups:
- Part A: Palovarotene 10/5 mg - Flare-up: Participants received palovarotene 10 mg for 14 days followed by 5 mg for 28 days during flare-ups (10/5-mg regimen). The participants were followed for an additional 42 days without treatment.
- Part B: Flare-up Combined: Skeletally mature participants received palovarotene 20 mg for 28 days followed by 10 mg for 56 days during flare-ups (20/10-mg regimen) and 5 mg daily when not taking flare-up dosing. Treatment may have been extended if the flare-up was ongoing and continued until the flare-up resolved. Dosing was extended in 4-week intervals and was based on clinical signs and symptoms as assessed by the Investigator.
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Flare-ups) | 28 | 51
percentage of flare-ups | 64.3 | 72.5

2. Primary Outcome: Parts B and C: Annualized Change in New HO Volume
Description: The annualized change in new HO volume was assessed by low-dose whole body computed tomography (WBCT) scan, excluding head. Results are presented for overall intent to treat (ITT) period.
Time Frame: From Baseline (Day 1) up to end of 2 year follow-up period, approximately a maximum of 96 months
Population: The Full Analysis Set (FAS) included all enrolled participants having a baseline HO volume measurement and at least 1 post-baseline HO volume measurement in the PVO-1A-202 study.
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)/year
Groups:
- Part B: Palovarotene - All Treated Flare-ups: Participants received palovarotene 20 mg for 28 days followed by 10 mg for 56 days during flare-ups and with 5 mg daily when not taking flare-up dosing for skeletally mature participants. Participants were treated for all flare-ups. The change in new HO total volume was compared to baseline where the baseline value was performed prior to the initiation of non-flare-up based dosing (in Part B).
- Part B: Untreated/Undertreated Flare-ups: Participants received palovarotene 20 mg for 28 days followed by 10 mg for 56 days during flare-ups and with 5 mg daily when not taking flare-up dosing for skeletally mature participants. At least 1 flare-up was untreated/undertreated. The change in new HO total volume was compared to baseline where the baseline value was performed prior to the initiation of non-flare-up based dosing (in Part B).
- Part B: No Flare-ups: Participants received palovarotene 5 mg daily. No flare-ups were reported. The change in new HO total volume was compared to baseline where the baseline value was performed prior to the initiation of non-flare-up based dosing (in Part B).
- Part B: All Treated and No Flare-ups Combined: Participants received palovarotene 20 mg for 28 days followed by 10 mg for 56 days during flare-ups and with 5 mg daily when not taking flare-up dosing for skeletally mature participants. This group pools data from all participants irrespective of treatment. The change in new HO total volume was compared to baseline where the baseline value was performed prior to the initiation of non-flare-up based dosing (in Part B).
- Part C: Palovarotene - All Treated Flare-ups: Participants received palovarotene 5 mg daily and 20 mg for 28 days followed by 10 mg for 56 days during flare-ups. Participants were treated for all flare-ups. The change in new HO total volume was compared to baseline where the baseline value was performed prior to the initiation of non-flare-up based dosing (in Part B or Part C).
- Part C: Untreated/Undertreated Flare-ups: At least 1 flare-up was untreated/undertreated. The change in new HO total volume was compared to baseline where the baseline value was performed prior to the initiation of non-flare-up based dosing (in Part B or Part C).
- Part C: No Flare-ups: No flare-ups were reported. The change in new HO total volume was compared to baseline where the baseline value was performed prior to the initiation of non-flare-up based dosing (in Part B or Part C).
- Part C: All Treated and No Flare-ups Combined: This group pools data from all participants irrespective of treatment. The change in new HO total volume was compared to baseline where the baseline value was performed prior to the initiation of non-flare-up based dosing (in Part B or Part C).
Arm/Group | Part B: Palovarotene - All Treated Flare-ups | Part B: Untreated/Undertreated Flare-ups | Part B: No Flare-ups | Part B: All Treated and No Flare-ups Combined | Part C: Palovarotene - All Treated Flare-ups | Part C: Untreated/Undertreated Flare-ups | Part C: No Flare-ups | Part C: All Treated and No Flare-ups Combined
Number analyzed (Participants) | 4 | 24 | 9 | 13 | 8 | 6 | 7 | 15
cubic millimeter (mm^3)/year | -3464.0 (5081.50) | 29522.8 (89408.15) | 25041.1 (58529.79) | 16270.3 (49777.40) | -10343.4 (18007.89) | 52291.4 (86019.62) | 30530.9 (51800.47) | 8731.3 (41924.30)

3. Secondary Outcome: Parts A and B: Percentage of Participants Across the 7 HO Scores at Month 12 of Part A; and Weeks 6 and 12 for Part B
Description: The HO score ranged from 0 to 6 where, 0 = no HO and 6 = single contiguous HO with longest dimension >2 diameters of the reference normotopic bone in any projection. Highest HO score from 2 projections was used.
Time Frame: Part A: Baseline (pre-dose data from Study PVO-1A-201 for follow-up component and flare-up screening/Day 1 for flare-up component) and Month 12; Part B: Baseline (flare-up screening/baseline) and Weeks 6 and 12
Population: No participants were analyzed for this endpoint.
Groups:
- Part B: Flare-up Combined: Participants received palovarotene 20 mg for 28 days followed by 10 mg for 56 days during flare-ups (20/10-mg regimen) and with 5 mg daily when not taking flare-up dosing for skeletally mature participants. Treatment may have been extended if the flare-up was ongoing and continued until the flare-up resolved. Dosing was extended in 4-week intervals and was based on clinical signs and symptoms as assessed by the Investigator.
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Parts A and B: Volume of New Heterotopic Bone Formed at Month 12
Description: Plain radiographs were utilized in Part A of the study. The interpretation of radiographs was to have documented the absence or presence of new HO at the flare-up site compared with the baseline assessment, and the volume of new HO if present. Low-dose CT scans were utilized in Part B of the study. Low-dose, flare-up site-specific CT scan was used as the primary imaging assessment of HO for flare-ups and low-dose, WBCT scans were used as the primary imaging assessment for total body HO in those participants receiving chronic treatment.
Time Frame: Month 12
Population: Part A: The Efficacy population included all participants in the treated population who had an evaluable Week 6 or Week 12 image (CT scan or plain radiograph).
  Part B: The Flare-up population included all participants in the treated population who took at least 1 dose of palovarotene during flare-up based treatment in Part B. Only participants with flare-ups at Week 12 are reported.
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 26 | 48
mm^3 | 2310 (4739) | 4818 (17349)

5. Secondary Outcome: Parts A and B: Number of Flare-ups With Significant Abnormalities in Cartilage, Bone, Angiogenesis, and Inflammation Biomarkers at Week 12
Description: Blood and urine samples for cartilage, bone, angiogenesis, and inflammation biomarkers were evaluated during Part A and Part B of the study. Bone and cartilage biomarkers included: osteocalcin, bone-specific alkaline phosphatase (ALP), procollagen type 1-N-terminal pro-peptide (PINP), cartilage-derived (CD) retinoic acid protein, procollagen type 1-C-terminal pro-peptide (PICP), and C-terminal telopeptide. Angiogenesis included urinary basic fibroblast growth factor. Inflammation included erythrocyte sedimentation rate, C-reactive protein, Interleukin(IL)-6, IL-1 beta, tumor necrosis factor (TNF)-alpha, creatine phosphokinase, and lactate dehydrogenase. Based on emerging data from studies PVO-1A-001, PVO-1A-201, and Parts A and B of PVO-1A-202, biomarkers were removed from the evaluation during Part C.
Time Frame: Part A and B: At Week 12
Population: Part A: The Efficacy population. Part B: The Flare-up population. The data collected for flare-ups used each flare-up as the unit of analysis rather than each participant. Additionally, a study participant may have not had any flare-ups whereas another participant may have had multiple flare-ups (note, the number of flare-ups can be larger than the number of participants OR it can be smaller OR it can match, by chance).
Measure: Number; unit: number of flare-ups
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 26 | 46
number of flare-ups
  Parts A and B: Osteocalcin: number analyzed (Participants) | 20 | 31
  Parts A and B: Osteocalcin: number analyzed (Number of flare-ups) | 25 | 44
  Parts A and B: Osteocalcin | 10 | 6
  Parts A and B: Bone-specific ALP: number analyzed (Participants) | 20 | 32
  Parts A and B: Bone-specific ALP: number analyzed (Number of flare-ups) | 26 | 45
  Parts A and B: Bone-specific ALP | 2 | 2
  Parts A and B: P1NP: number analyzed (Participants) | 20 | 31
  Parts A and B: P1NP: number analyzed (Number of flare-ups) | 25 | 44
  Parts A and B: P1NP | 10 | 2
  Parts A and B: CD retinoic acid protein: number analyzed (Participants) | 20 | 32
  Parts A and B: CD retinoic acid protein: number analyzed (Number of flare-ups) | 26 | 45
  Parts A and B: CD retinoic acid protein | 4 | 6
  Parts A and B: P1CP: number analyzed (Participants) | 20 | 32
  Parts A and B: P1CP | 3 | 2
  Parts A and B: C-terminal telopeptide: number analyzed (Participants) | 20 | 32
  Parts A and B: C-terminal telopeptide | 0 | 1
  Parts A and B: Urinary basic FGF: number analyzed (Participants) | 17 | 32
  Parts A and B: Urinary basic FGF: number analyzed (Number of flare-ups) | 23 | 43
  Parts A and B: Urinary basic FGF | 6 | 5
  Parts A and B: ESR: number analyzed (Participants) | 19 | 32
  Parts A and B: ESR: number analyzed (Number of flare-ups) | 26 | 43
  Parts A and B: ESR | 4 | 0
  Parts A and B: C-reactive protein: number analyzed (Participants) | 20 | 29
  Parts A and B: C-reactive protein: number analyzed (Number of flare-ups) | 24 | 43
  Parts A and B: C-reactive protein | 6 | 5
  Parts A and B: IL-6: number analyzed (Participants) | 20 | 32
  Parts A and B: IL-6 | 0 | 3
  Parts A and B: IL-1 beta: number analyzed (Participants) | 20 | 32
  Parts A and B: IL-1 beta | 5 | 5
  Parts A and B: TNF-alpha: number analyzed (Participants) | 20 | 32
  Parts A and B: TNF-alpha | 3 | 1
  Parts A and B: Creatine kinase: number analyzed (Participants) | 20 | 29
  Parts A and B: Creatine kinase: number analyzed (Number of flare-ups) | 24 | 43
  Parts A and B: Creatine kinase | 1 | 3
  Parts A and B: Lactate dehydrogenase: number analyzed (Participants) | 20 | 29
  Parts A and B: Lactate dehydrogenase: number analyzed (Number of flare-ups) | 24 | 42
  Parts A and B: Lactate dehydrogenase | 4 | 1

6. Secondary Outcome: Parts A and B: Change From Baseline in Active Range of Motion (ROM) at Flare-up Site at Week 12
Description: Active ROM was assessed by goniometer in Parts A and B of the study. Measurements were performed by trained and qualified study personnel (eg, physiotherapist) in order to standardize the performance of procedures and minimize variability. Flare-ups at the primary joint was expressed as percent of normal arc of motion. Based on the change in the schedule for flare-up based assessments. Baseline was defined as pre-dose data from Study PVO-1A-201 for follow-up component and flare-up screening/Day 1 for flare-up component for Part A and flare-up screening/baseline for Part B.
Time Frame: Baseline and Week 12
Population: Part A: Efficacy population included all participants in the treated population who had an evaluable Week 6 or Week 12 image (CT scan or plain radiograph).
  Part B: Flare-up population included all participants in the treated population who took at least 1 dose of palovarotene during flare-up based treatment in Part B. Only participants with flare-ups at baseline and Week 12 are reported.
Measure: Mean (Standard Deviation); unit: percent of normal total arc of motion
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 27 | 49
percent of normal total arc of motion | -6.16 (14.362) | -0.49 (18.096)

7. Secondary Outcome: Part B: Change From Baseline in ROM at Week 12
Description: The ROM was assessed by the Investigator using Cumulative Analogue Joint Involvement Scale (CAJIS) for participants in Part B. It includes 12 joints (shoulder, elbow, wrist, hip, knee, and ankle on both the right and left sides), and 3 body regions (jaw, cervical spine [neck], and thoracic/lumbar spine). Each joint/region was assessed as: 0=uninvolved; 1=partially involved; and 2=completely ankylosed. The total score range is 0 (no involvement) to 30 (maximally involved). Baseline was flare-up screening.
Time Frame: Baseline and Week 12
Population: Flare-up population. The data collected for flare-ups used each flare-up as unit of analysis rather than each participant. Additionally, a study participant may have not had any flare-ups whereas another participant may have had multiple flare-ups (note, the number of flare-ups can be larger than the number of participants OR it can be smaller OR it can match, by chance). Only participants with flare-ups at baseline and at each time point are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of flare-ups
Arm/Group | Part B: Flare-up Combined
Number analyzed (Participants) | 33
Number analyzed (Number of flare-ups) | 51
units on a scale | 0.3 (1.80)

8. Secondary Outcome: Part C: Change From Baseline in ROM at Months 6, 12, 18, 24, 30, 36, 42, and 48
Description: The ROM was assessed by the Investigator using CAJIS for participants in Part C. It includes 12 joints (shoulder, elbow, wrist, hip, knee, and ankle on both the right and left sides), and 3 body regions (jaw, cervical spine [neck], and thoracic/lumbar spine). Each joint/region was assessed as: 0=uninvolved; 1=partially involved; and 2=completely ankylosed. The total score range is 0 (no involvement) to 30 (maximally involved). Baseline was chronic Day 1.
Time Frame: Baseline and Months 6, 12, 18, 24, 30, 36, 42, and 48
Population: The Safety analysis set included all enrolled participants who received at least 1 dose of palovarotene in the PVO-1A-202 study. Only participants analyzed at baseline and specific time point are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part C: Palovarotene - All Treated Flare-ups
Number analyzed (Participants) | 34
units on a scale
  Month 6: number analyzed (Participants) | 31
  Month 6 | 0.2 (1.58)
  Month 12 | 0.6 (1.76)
  Month 18: number analyzed (Participants) | 26
  Month 18 | 0.9 (1.73)
  Month 24: number analyzed (Participants) | 31
  Month 24 | 1.3 (2.74)
  Month 30: number analyzed (Participants) | 26
  Month 30 | 1.5 (2.79)
  Month 36: number analyzed (Participants) | 25
  Month 36 | 1.6 (3.38)
  Month 42: number analyzed (Participants) | 23
  Month 42 | 1.6 (3.03)
  Month 48: number analyzed (Participants) | 5
  Month 48 | 3.0 (2.55)

9. Secondary Outcome: Part B: Participant and Investigator Global Assessment of Movement at Week 12
Description: Participants/Investigators assessed how the flare-up was affecting movement (better, same, slightly worse, moderately worse, or severely worse movement) compared with baseline. Based on the change in the schedule for flare-up based assessments. PA = Participant assessment and IA = Investigator assessment.
Time Frame: Week 12
Population: The Flare-up population. The data collected for flare-ups used each flare-up as the unit of analysis rather than each participant. Additionally, a study participant may have not had any flare-ups whereas another participant may have had multiple flare-ups (note, the number of flare-ups can be larger than the number of participants OR it can be smaller OR it can match, by chance). Only participants with flare-ups at baseline and Week 12 are reported.
Measure: Number; unit: number of flare-ups
Units Other Than Participants: Flare-ups
Arm/Group | Part B: Flare-up Combined
Number analyzed (Participants) | 35
Number analyzed (Flare-ups) | 51
number of flare-ups
  PA: New HO - Better movement: number analyzed (Participants) | 12
  PA: New HO - Better movement: number analyzed (Flare-ups) | 14
  PA: New HO - Better movement | 5
  PA: New HO - Same movement: number analyzed (Participants) | 12
  PA: New HO - Same movement: number analyzed (Flare-ups) | 14
  PA: New HO - Same movement | 3
  PA: New HO - Slightly worse movement: number analyzed (Participants) | 12
  PA: New HO - Slightly worse movement: number analyzed (Flare-ups) | 14
  PA: New HO - Slightly worse movement | 2
  PA: New HO - Moderately worse movement: number analyzed (Participants) | 12
  PA: New HO - Moderately worse movement: number analyzed (Flare-ups) | 14
  PA: New HO - Moderately worse movement | 2
  PA: New HO - Severely worse movement: number analyzed (Participants) | 12
  PA: New HO - Severely worse movement: number analyzed (Flare-ups) | 14
  PA: New HO - Severely worse movement | 2
  PA: No new HO - Better movement: number analyzed (Participants) | 23
  PA: No new HO - Better movement: number analyzed (Flare-ups) | 37
  PA: No new HO - Better movement | 11
  PA: No new HO - Same movement: number analyzed (Participants) | 23
  PA: No new HO - Same movement: number analyzed (Flare-ups) | 37
  PA: No new HO - Same movement | 20
  PA: No new HO - Slightly worse movement: number analyzed (Participants) | 23
  PA: No new HO - Slightly worse movement: number analyzed (Flare-ups) | 37
  PA: No new HO - Slightly worse movement | 5
  PA: No new HO - Moderately worse movement: number analyzed (Participants) | 23
  PA: No new HO - Moderately worse movement: number analyzed (Flare-ups) | 37
  PA: No new HO - Moderately worse movement | 1
  PA: No new HO - Severely worse movement: number analyzed (Participants) | 23
  PA: No new HO - Severely worse movement: number analyzed (Flare-ups) | 37
  PA: No new HO - Severely worse movement | 0
  IA: New HO - Better movement: number analyzed (Participants) | 12
  IA: New HO - Better movement: number analyzed (Flare-ups) | 14
  IA: New HO - Better movement | 5
  IA: New HO - Same movement: number analyzed (Participants) | 12
  IA: New HO - Same movement: number analyzed (Flare-ups) | 14
  IA: New HO - Same movement | 3
  IA: New HO - Slightly worse movement: number analyzed (Participants) | 12
  IA: New HO - Slightly worse movement: number analyzed (Flare-ups) | 14
  IA: New HO - Slightly worse movement | 2
  IA: New HO - Moderately worse movement: number analyzed (Participants) | 12
  IA: New HO - Moderately worse movement: number analyzed (Flare-ups) | 14
  IA: New HO - Moderately worse movement | 3
  IA: New HO - Severely worse movement: number analyzed (Participants) | 12
  IA: New HO - Severely worse movement: number analyzed (Flare-ups) | 14
  IA: New HO - Severely worse movement | 1
  IA: No new HO - Better movement: number analyzed (Participants) | 23
  IA: No new HO - Better movement: number analyzed (Flare-ups) | 37
  IA: No new HO - Better movement | 1
  IA: No new HO - Same movement: number analyzed (Participants) | 23
  IA: No new HO - Same movement: number analyzed (Flare-ups) | 37
  IA: No new HO - Same movement | 29
  IA: No new HO - Slightly worse movement: number analyzed (Participants) | 23
  IA: No new HO - Slightly worse movement: number analyzed (Flare-ups) | 37
  IA: No new HO - Slightly worse movement | 6
  IA: No new HO - Moderately worse movement: number analyzed (Participants) | 23
  IA: No new HO - Moderately worse movement: number analyzed (Flare-ups) | 37
  IA: No new HO - Moderately worse movement | 1
  IA: No new HO - Severely worse movement: number analyzed (Participants) | 23
  IA: No new HO - Severely worse movement: number analyzed (Flare-ups) | 37
  IA: No new HO - Severely worse movement | 0

10. Secondary Outcome: Part A: Change From Baseline in Numeric Rating Scale (NRS) Pain and Swelling or Faces Pain Scale-Revised (FPS-R) at Weeks 2, 4, 6, 9, and 12
Description: The NRSs for pain and swelling were used in Part A of the study to evaluate the effect of palovarotene on pain and swelling at the flare-up site. Flare-up pain was rated on a scale ranging from 0 (no pain or swelling) to 10 (worst pain or swelling ever experienced). For children less than 8 years old, pain was rated using the FPS-R, which ranging from 0 to 10 in 2-point increments where 0 = no pain and 10 = very much pain. Flare-up swelling was rated on a scale from 0 to 10 where 0 = no swelling and 10 = worst swelling ever experienced. Higher scores indicate worst quality of life for all scales. Baseline was predose data from PVO-1A-201 study/flare-up screening/Day 1.
Time Frame: Baseline and Weeks 2, 4, 6, 9, and 12
Population: The Efficacy population. The data collected for flare-ups used each flare-up as unit of analysis rather than each participant. Additionally, a study participant may have not had any flare-ups whereas another participant may have had multiple flare-ups (note, number of flare-ups can be larger than the number of participants OR it can be smaller OR it can match, by chance). Only participants with flare-ups at baseline and at each time point are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up
Number analyzed (Participants) | 20
Number analyzed (Number of flare-ups) | 28
units on a scale
  Week 2: Pain: number analyzed (Number of flare-ups) | 27
  Week 2: Pain | -1.4 (2.22)
  Week 4: Pain | -2.1 (2.27)
  Week 6: Pain | -2.6 (2.71)
  Week 9: Pain: number analyzed (Participants) | 15
  Week 9: Pain: number analyzed (Number of flare-ups) | 18
  Week 9: Pain | -2.9 (2.97)
  Week 12: Pain | -2.6 (2.85)
  Week 2: Swelling: number analyzed (Number of flare-ups) | 27
  Week 2: Swelling | -1.7 (1.83)
  Week 4: Swelling | -2.3 (2.31)
  Week 6: Swelling | -2.4 (2.38)
  Week 9: Swelling: number analyzed (Participants) | 15
  Week 9: Swelling: number analyzed (Number of flare-ups) | 18
  Week 9: Swelling | -2.7 (2.47)
  Week 12: Swelling | -2.9 (2.46)

11. Secondary Outcome: Parts A and B: Change From Baseline in Physical Function at Weeks 2, 4, 6, 9, and 12 of Part A; and Weeks 4, 8, and 12 of Part B
Description: The effect of palovarotene on physical function was determined using Fibrodysplasia Ossificans Progressiva-Physical Function Questionnaire (FOP-PFQ). The questionnaire consisted of 28 items ranging from 1 (not able to do) to 5 (with no trouble; without help or assistive device). Total score range from 28 to 140. Lower scores denoted more difficulty, with items categorized into upper extremity and mobility sections.
Time Frame: Part A: Baseline and Weeks 2, 4, 6, 9, and 12; and Part B: Baseline and Weeks 4, 8, and 12
Population: Part A: Efficacy population. Part B: Flare-up population. Data collected for flare-ups used each flare-up as unit of analysis rather than each participant. A study participant may have not had any flare-ups whereas another participant may have had multiple flare-ups (number of flare-ups can be larger than number of participants OR it can be smaller OR it can match, by chance). Only participants with flare-ups at baseline and at each time point are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 28 | 52
units on a scale
  Parts A and B: Week 2: number analyzed (Participants) | 20 | 0
  Parts A and B: Week 2: number analyzed (Number of flare-ups) | 27 | 0
  Parts A and B: Week 2 | -0.97 (4.939) |
  Parts A and B: Week 4: number analyzed (Participants) | 20 | 29
  Parts A and B: Week 4: number analyzed (Number of flare-ups) | 28 | 47
  Parts A and B: Week 4 | 0.38 (4.746) | -1.23 (4.453)
  Parts A and B: Week 6: number analyzed (Participants) | 20 | 0
  Parts A and B: Week 6: number analyzed (Number of flare-ups) | 28 | 0
  Parts A and B: Week 6 | 0.21 (6.501) |
  Parts A and B: Week 8: number analyzed (Participants) | 0 | 32
  Parts A and B: Week 8: number analyzed (Number of flare-ups) | 0 | 50
  Parts A and B: Week 8 |  | 0.88 (9.357)
  Parts A and B: Week 9: number analyzed (Participants) | 15 | 0
  Parts A and B: Week 9: number analyzed (Number of flare-ups) | 18 | 0
  Parts A and B: Week 9 | 0.76 (6.054) |
  Parts A and B: Week 12: number analyzed (Participants) | 20 | 32
  Parts A and B: Week 12: number analyzed (Number of flare-ups) | 28 | 50
  Parts A and B: Week 12 | 0.69 (6.604) | 0.17 (6.893)

12. Secondary Outcome: Part C: Change From Baseline in Physical Function at Months 6, 12, 18, 24, 30, 36, 42, and 48
Description: The effect of palovarotene on physical function was determined using FOP-PFQ. The questionnaire consisted of 28 items ranging from 1 (not able to do) to 5 (with no trouble; without help or assistive device). Total score range from 28 to 140. Lower scores denoted more difficulty, with items categorized into upper extremity and mobility sections.
Time Frame: Baseline and Months 6, 12, 18, 24, 30, 36, 42, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part C: Palovarotene - All Treated Flare-ups
Number analyzed (Participants) | 36
units on a scale
  Month 6 | 1.8 (6.36)
  Month 12 | 1.8 (9.81)
  Month 18: number analyzed (Participants) | 31
  Month 18 | 4.0 (9.49)
  Month 24: number analyzed (Participants) | 31
  Month 24 | 7.5 (14.00)
  Month 30: number analyzed (Participants) | 27
  Month 30 | 8.2 (13.45)
  Month 36: number analyzed (Participants) | 24
  Month 36 | 9.8 (14.11)
  Month 42: number analyzed (Participants) | 22
  Month 42 | 7.0 (13.14)
  Month 48: number analyzed (Participants) | 7
  Month 48 | 8.3 (7.76)

13. Secondary Outcome: Parts A and B: Change From Baseline in Physical and Mental Health at Weeks 2, 4, 6, 9, and 12 of Part A; and Weeks 4, 8, and 12 of Part B
Description: The patient reported outcomes measurement information system (PROMIS) global health scale was administered to evaluate the effect of palovarotene on physical and mental health in participants ≥15 years of age and mental health in participants <15 years of age, age-appropriate forms of the PROMIS global health scales were administered. A T-score of 50 is normal and increments of 10 are +/- standard deviation away from the norm. A T-score <50 indicates worse health, while a T-score >50 indicates better health. Higher values (positive changes) indicate better health. AFPH = Adult Form, Physical Health; AFMH = Adult Form, Mental Health; PFH = Paediatric Form, Health.
Time Frame: Part A: Baseline and Weeks 2, 4, 6, 9, and 12; and Part B: Baseline and Weeks 4, 8, and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 28 | 52
units on a scale
  Parts A and B: AFPH - Week 2: number analyzed (Participants) | 18 | 0
  Parts A and B: AFPH - Week 2: number analyzed (Number of flare-ups) | 25 | 0
  Parts A and B: AFPH - Week 2 | 3.26 (4.819) |
  Parts A and B: AFPH - Week 4: number analyzed (Participants) | 18 | 20
  Parts A and B: AFPH - Week 4: number analyzed (Number of flare-ups) | 26 | 32
  Parts A and B: AFPH - Week 4 | 2.14 (3.976) | 0.2 (3.17)
  Parts A and B: AFPH - Week 6: number analyzed (Participants) | 18 | 0
  Parts A and B: AFPH - Week 6: number analyzed (Number of flare-ups) | 26 | 0
  Parts A and B: AFPH - Week 6 | 1.78 (3.735) |
  Parts A and B: AFPH - Week 8: number analyzed (Participants) | 0 | 21
  Parts A and B: AFPH - Week 8: number analyzed (Number of flare-ups) | 0 | 33
  Parts A and B: AFPH - Week 8 |  | 0.3 (3.33)
  Parts A and B: AFPH - Week 9: number analyzed (Participants) | 13 | 0
  Parts A and B: AFPH - Week 9: number analyzed (Number of flare-ups) | 16 | 0
  Parts A and B: AFPH - Week 9 | 2.87 (5.352) |
  Parts A and B: AFPH - Week 12: number analyzed (Participants) | 18 | 22
  Parts A and B: AFPH - Week 12: number analyzed (Number of flare-ups) | 26 | 34
  Parts A and B: AFPH - Week 12 | 3.22 (4.855) | 0.6 (3.79)
  Parts A and B: AFMH - Week 2: number analyzed (Participants) | 18 | 0
  Parts A and B: AFMH - Week 2: number analyzed (Number of flare-ups) | 25 | 0
  Parts A and B: AFMH - Week 2 | 1.00 (4.667) |
  Parts A and B: AFMH - Week 4: number analyzed (Participants) | 18 | 20
  Parts A and B: AFMH - Week 4: number analyzed (Number of flare-ups) | 26 | 32
  Parts A and B: AFMH - Week 4 | 0.39 (3.264) | 1.0 (8.05)
  Parts A and B: AFMH - Week 6: number analyzed (Participants) | 18 | 0
  Parts A and B: AFMH - Week 6: number analyzed (Number of flare-ups) | 26 | 0
  Parts A and B: AFMH - Week 6 | 1.03 (3.122) |
  Parts A and B: AFMH - Week 8: number analyzed (Participants) | 0 | 21
  Parts A and B: AFMH - Week 8: number analyzed (Number of flare-ups) | 0 | 33
  Parts A and B: AFMH - Week 8 |  | -0.3 (7.47)
  Parts A and B: AFMH - Week 9: number analyzed (Participants) | 13 | 0
  Parts A and B: AFMH - Week 9: number analyzed (Number of flare-ups) | 16 | 0
  Parts A and B: AFMH - Week 9 | -0.16 (4.422) |
  Parts A and B: AFMH - Week 12: number analyzed (Participants) | 18 | 22
  Parts A and B: AFMH - Week 12: number analyzed (Number of flare-ups) | 26 | 34
  Parts A and B: AFMH - Week 12 | 0.99 (2.915) | 0.2 (7.63)
  Parts A and B: PFH - Week 2: number analyzed (Participants) | 2 | 0
  Parts A and B: PFH - Week 2: number analyzed (Number of flare-ups) | 2 | 0
  Parts A and B: PFH - Week 2 | -0.05 (2.475) |
  Parts A and B: PFH - Week 4: number analyzed (Participants) | 2 | 10
  Parts A and B: PFH - Week 4: number analyzed (Number of flare-ups) | 2 | 16
  Parts A and B: PFH - Week 4 | 1.70 (4.950) | 0.7 (4.77)
  Parts A and B: PFH - Week 6: number analyzed (Participants) | 2 | 0
  Parts A and B: PFH - Week 6: number analyzed (Number of flare-ups) | 2 | 0
  Parts A and B: PFH - Week 6 | 5.25 (4.596) |
  Parts A and B: PFH - Week 8: number analyzed (Participants) | 0 | 10
  Parts A and B: PFH - Week 8: number analyzed (Number of flare-ups) | 0 | 16
  Parts A and B: PFH - Week 8 |  | -2.5 (6.32)
  Parts A and B: PFH - Week 9: number analyzed (Participants) | 2 | 0
  Parts A and B: PFH - Week 9: number analyzed (Number of flare-ups) | 2 | 0
  Parts A and B: PFH - Week 9 | 0.85 (1.202) |
  Parts A and B: PFH - Week 12: number analyzed (Participants) | 2 | 10
  Parts A and B: PFH - Week 12: number analyzed (Number of flare-ups) | 2 | 16
  Parts A and B: PFH - Week 12 | 0.85 (3.748) | 0.4 (5.65)

14. Secondary Outcome: Part C: Change From Baseline in Physical and Mental Health at Months 6, 12, 18, 24, 30, 36, 42, and 48
Description: The PROMIS global health scale was administered to evaluate the effect of palovarotene on physical and mental health in participants ≥15 years of age and mental health in participants <15 years of age, age-appropriate forms of the PROMIS global health scales were administered. A T-score of 50 is normal and increments of 10 are +/- standard deviation away from the norm. A T-score <50 indicates worse health, while a T-score >50 indicates better health. Higher values (positive changes) indicate better health. AFPH = Adult Form, Physical Health; AFMH = Adult Form, Mental Health; PFH = Paediatric Form, Health.
Time Frame: Baseline and Months 6, 12, 18, 24, 30, 36, 42, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part C: Palovarotene - All Treated Flare-ups
Number analyzed (Participants) | 30
units on a scale
  AFPH - Month 6 | -0.2 (5.59)
  AFPH - Month 12 | 0.6 (6.04)
  AFPH - Month 18: number analyzed (Participants) | 24
  AFPH - Month 18 | -0.1 (5.30)
  AFPH - Month 24: number analyzed (Participants) | 25
  AFPH - Month 24 | -1.1 (7.10)
  AFPH - Month 30: number analyzed (Participants) | 22
  AFPH - Month 30 | 0.1 (4.46)
  AFPH - Month 36: number analyzed (Participants) | 22
  AFPH - Month 36 | -1.1 (5.97)
  AFPH - Month 42: number analyzed (Participants) | 21
  AFPH - Month 42 | -1.8 (6.55)
  AFPH - Month 48: number analyzed (Participants) | 5
  AFPH - Month 48 | -1.6 (3.02)
  AFMH - Month 6 | -2.2 (6.49)
  AFMH - Month 12 | -0.0 (3.96)
  AFMH - Month 18: number analyzed (Participants) | 25
  AFMH - Month 18 | -0.8 (5.04)
  AFMH - Month 24: number analyzed (Participants) | 25
  AFMH - Month 24 | -2.5 (5.96)
  AFMH - Month 30: number analyzed (Participants) | 22
  AFMH - Month 30 | -3.0 (5.30)
  AFMH - Month 36: number analyzed (Participants) | 22
  AFMH - Month 36 | -1.5 (4.95)
  AFMH - Month 42: number analyzed (Participants) | 21
  AFMH - Month 42 | -2.9 (6.24)
  AFMH - Month 48: number analyzed (Participants) | 6
  AFMH - Month 48 | -5.2 (7.83)
  PFH - Month 6: number analyzed (Participants) | 4
  PFH - Month 6 | 3.8 (2.91)
  PFH - Month 12: number analyzed (Participants) | 3
  PFH - Month 12 | 1.7 (1.65)
  PFH - Month 18: number analyzed (Participants) | 3
  PFH - Month 18 | 4.7 (1.93)
  PFH - Month 24: number analyzed (Participants) | 3
  PFH - Month 24 | 3.4 (4.63)
  PFH - Month 30: number analyzed (Participants) | 3
  PFH - Month 30 | 4.6 (2.52)

15. Secondary Outcome: Parts A and B: Number of Any Assistive Devices and Adaptations by FOP Participants at Weeks 6 and 12 of Part A; and Week 12 of Part B
Description: The FOP assistive devices and adaptations questionnaire was used in Part A and Part B of the study. Assistive devices and adaptations were grouped into the following categories: mobility aids, care attendants, eating tools, personal care tools/aids, bathroom aids and devices, bedroom aids and devices, home adaptations, work environment adaptations, technology adaptations, sports and recreation adaptations, school, and medical therapies for daily living. When a flare-up did not use an assistive device or adaptation or considered the assistive device or adaptation not applicable, 0 was imputed for analysis.
Time Frame: Part A: Weeks 6 and 12; and Part B: Week 12
Population: Part A: The Efficacy population. Part B: The Flare-up population. Only participants with flare-ups at baseline and at each time point are reported.
Measure: Mean (Standard Deviation); unit: devices adaptations
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 28 | 52
devices adaptations
  Part A: Week 6: number analyzed (Participants) | 20 | 0
  Part A: Week 6: number analyzed (Number of flare-ups) | 28 | 0
  Part A: Week 6 | 12.9 (11.52) |
  Parts A and B: Week 12 | 14.3 (12.39) | 13.2 (10.50)

16. Secondary Outcome: Part A: Percentage of Responders at Week 12
Description: A responder was defined as a participant with no or minimal new HO at original flare-up site compared with baseline (flare-up screening/Day 1). Minimal new HO was defined as new HO with an HO score <=3 in both the AP and lateral projections (or if 1 view is non-interpretable or non-evaluable, then remaining evaluable view was used). The HO score ranged from 0 to 6 where, 0 = no HO and 6 = single contiguous HO with longest dimension >2 diameters of the reference normotopic bone in any projection. Highest HO score from 2 projections was used. Results from the Primary Read reviews are presented.
Time Frame: Week 12
Population: The Efficacy population included all participants in the treated population who had an evaluable Week 6 or Week 12 image (CT scan or plain radiograph). Only participants with flare-ups at baseline and Week 12 are reported.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up
Number analyzed (Participants) | 20
Number analyzed (Number of flare-ups) | 28
percentage of participants | 64.3

17. Secondary Outcome: Parts A and B: Change From Baseline in Amount of Bone Formation Biomarker at Weeks 6 and 12 of Part A; and Week 12 of Part B
Description: The bone formation was measured by PINP biomarker. Baseline was defined as flare-up screening/Day 1.
Time Frame: Part A: Baseline and Weeks 6 and 12; and Part B: Baseline and Week 12
Population: Part A: The Efficacy population. Part B: The Flare-up population. The data collected for flare-ups used each flare-up as unit of analysis rather than each participant. Additionally, a study participant may have not had any flare-ups whereas another participant may have had multiple flare-ups (note, number of flare-ups can be larger than the number of participants OR it can be smaller OR it can match, by chance). Only participants with flare-ups at baseline and at each time point are reported.
Measure: Mean (Standard Deviation); unit: microgram per liter
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 28 | 52
microgram per liter
  Part A: Week 6: number analyzed (Participants) | 14 | 0
  Part A: Week 6: number analyzed (Number of flare-ups) | 18 | 0
  Part A: Week 6 | 38.755 (50.547) |
  Parts A and B: Week 12: number analyzed (Participants) | 15 | 27
  Parts A and B: Week 12: number analyzed (Number of flare-ups) | 18 | 39
  Parts A and B: Week 12 | 54.592 (140.540) | 70.916 (130.608)

18. Secondary Outcome: Parts A and B: Number of Flare-ups With Soft Tissue Swelling and/or Cartilage Formation at Weeks 6 and 12 of Part A; and Week 12 of Part B
Description: Magnetic resonance imaging (MRI) was utilized as an imaging modality to evaluate for the presence of soft tissue swelling/edema and cartilage formation for participants who received flare-up based treatment. Ultrasound (US) was utilized to evaluate for the presence of soft tissue swelling in participants unable to undergo MRI. Both MRI and US were interpreted centrally. When US was used, cartilage formation was not assessed.
Time Frame: Part A: Baseline and Weeks 6 and 12; and Part B: Baseline and Week 12
Population: as for outcome 17
Measure: Number; unit: flare-up
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 28 | 52
flare-up
  Part A: Edema - Week 6: number analyzed (Participants) | 14 | 0
  Part A: Edema - Week 6: number analyzed (Number of flare-ups) | 18 | 0
  Part A: Edema - Week 6 | 7 |
  Part A: Cartilage Formation - Week 6: number analyzed (Participants) | 10 | 0
  Part A: Cartilage Formation - Week 6: number analyzed (Number of flare-ups) | 12 | 0
  Part A: Cartilage Formation - Week 6 | 0 |
  Parts A and B: Edema - Week 12: number analyzed (Participants) | 13 | 32
  Parts A and B: Edema - Week 12: number analyzed (Number of flare-ups) | 17 | 49
  Parts A and B: Edema - Week 12 | 9 | 36
  Parts A and B: Cartilage Formation - Week 12: number analyzed (Participants) | 10 | 16
  Parts A and B: Cartilage Formation - Week 12: number analyzed (Number of flare-ups) | 12 | 22
  Parts A and B: Cartilage Formation - Week 12 | 0 | 1

19. Secondary Outcome: Parts A and B: Duration of Active Symptomatic Flare-up
Description: The number of days of active symptomatic flare-up was the number of days the participant reported the presence of symptoms in the diary.
Time Frame: Part A: From Baseline up to 36 months; and Part B: From Baseline up to 24 months
Population: Part A: The Efficacy population included all participants in the treated population who had an evaluable Week 6 or Week 12 image (CT scan or plain radiograph).
  Part B: The Flare-up population included all participants in the treated population who took at least 1 dose of palovarotene during flare-up based treatment in Part B. Only participants analyzed at baseline and specific time point are reported.
Measure: Mean (Standard Deviation); unit: day
Units Other Than Participants: Number of flare-ups
Arm/Group | Part A: Palovarotene 10/5 mg - Flare-up | Part B: Flare-up Combined
Number analyzed (Participants) | 20 | 35
Number analyzed (Number of flare-ups) | 24 | 48
day | 27.1 (29.9) | 39.5 (36.1)

20. Secondary Outcome: Part B: Change From Baseline in Whole Body Burden of HO at Months 12 and 24
Description: Whole body burden of HO was assessed by low-dose WBCT scan, excluding head. Baseline was Part B Screening.
Time Frame: Baseline and Months 12 and 24
Population: The WBCT Population included participants who received chronic dosing and had baseline and Month 12 WBCT scans. Only participants analyzed at baseline and specific time point are reported.
Measure: Mean (Standard Deviation); unit: mm^3
Groups:
- Part B: Whole Body Computed Tomography (WBCT) Population: Participants received palovarotene 20 mg for 28 days followed by 10 mg for 56 days during flare-ups (20/10-mg regimen) and with 5 mg daily when not taking flare-up dosing for skeletally mature participants. Treatment may have been extended if the flare-up was ongoing and continued until the flare-up resolved. Dosing was extended in 4-week intervals and was based on clinical signs and symptoms as assessed by the Investigator. The WBCT Population included participants who received chronic dosing and had Baseline and at least 1 post-baseline scan.
Arm/Group | Part B: Whole Body Computed Tomography (WBCT) Population
Number analyzed (Participants) | 37
mm^3
  Month 12: number analyzed (Participants) | 36
  Month 12 | 28386 (89918)
  Month 24: number analyzed (Participants) | 1
  Month 24 | 193150 (9999)

21. Secondary Outcome: Part B: Mean Percentage of Flare-ups Per Participant-Month Overall
Description: Flare-ups were counted using the number of participant/Investigator-reported flare-ups. Percentage was calculated by dividing the total number of flare-ups by the total participant months of follow-up. Results are presented for overall ITT period.
Time Frame: From Baseline (Day 1) up to end of 2 year follow-up period, approximately a maximum of 96 months
Population: The Safety analysis set included all enrolled participants who received at least 1 dose of palovarotene in the PVO-1A-202 study.
Measure: Mean (Standard Deviation); unit: percentage of flare-up/participant-month
Units Other Than Participants: Number of flare-ups
Arm/Group | Part B: Flare-up Combined
Number analyzed (Participants) | 35
Number analyzed (Number of flare-ups) | 52
percentage of flare-up/participant-month | 0.12 (0.124)

22. Secondary Outcome: Part C: Mean Percentage of Flare-ups Per Participant-Month Overall
Description: as for outcome 21
Time Frame: From Baseline (Day 1) up to end of 2 year follow-up period, approximately a maximum of 96 months
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage of flare-up/participant-month
Arm/Group | Part C: Palovarotene - All Treated Flare-ups
Number analyzed (Participants) | 46
percentage of flare-up/participant-month | 0.14 (0.150)

23. Secondary Outcome: Part C: Percentage of Participants With New HO at Months 12, 24, 36, 60, and 72 (Last Visit)
Description: New HO was defined as total WBCT new HO volume >0. Results for Month 72 are presented for overall ITT period.
Time Frame: Months 12, 24, 36, 60, and 72 (last visit)
Population: The FAS included all enrolled participants having a baseline HO volume measurement and at least 1 post-baseline HO volume measurement in the PVO-1A-202 study.
Measure: Number; unit: percentage of participants
Arm/Group | Part C: Palovarotene - All Treated Flare-ups
Number analyzed (Participants) | 46
percentage of participants
  Month 12: number analyzed (Participants) | 10
  Month 12 | 60.0
  Month 24: number analyzed (Participants) | 33
  Month 24 | 54.5
  Month 36: number analyzed (Participants) | 26
  Month 36 | 61.5
  Month 60: number analyzed (Participants) | 3
  Month 60 | 100.0
  Month 72: number analyzed (Participants) | 29
  Month 72 | 86.2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were recorded from the time informed consent was signed through end of the study (a maximum of 96 months).
Description: The Safety analysis set included all enrolled participants who received at least 1 dose of palovarotene in the PVO-1A-202 study.
Groups:
- Part A: Participants who completed PVO-1A-201 study were followed for up to 36 months in Part A. Eligible participants with a flare-up received palovarotene 10 mg capsule orally daily for 2 weeks followed by 5 mg daily for 4 weeks during the flare-up component of Part A.
- Part B: Eligible participants from Part A and participants from the new Adult Cohort received chronic treatment with palovarotene 5 mg daily for up to 24 months. Participants with flare-ups received palovarotene 20 mg daily for 4 weeks followed by 10 mg daily for 8 weeks.
- Part C: Eligible participants received chronic treatment of palovarotene 5 mg daily for up to 36 months. Participants with flare-ups received palovarotene 20mg daily for 4 weeks followed by 10 mg daily for 8 weeks. For skeletal immature participants, the exposure-equivalent dose was determined based on weight.
- Part D: Eligible participants were followed for up to an additional 48 months. No study drug was administered.
Arm/Group | Part A | Part B | Part C | Part D
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/52 | 0/46 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/20 | 9/52 | 25/46 | 0/1
Other Adverse Events (participants affected / at risk) | 20/20 | 52/52 | 46/46 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=20) | Part B (N=52) | Part C (N=46) | Part D (N=1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Condition aggravated (General disorders) | 1 (3) | 2 (4) | 2 (3) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (9) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epiphyses premature fusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (12) | 1 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=20) | Part B (N=52) | Part C (N=46) | Part D (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 6 (7) | 3 (3) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 4 (5) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 4 (5) | 12 (15) | 12 (13) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Eyelid skin dryness (Eye disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 3 (4) | 3 (3) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 4 (9) | 12 (12) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 5 (11) | 5 (6) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 2 (3) | 7 (14) | 4 (6) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 6 (6) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 8 (9) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 14 (19) | 8 (11) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 6 (7) | 8 (9) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 4 (9) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 9 (9) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 13 (17) | 32 (43) | 26 (31) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 15 (24) | 10 (17) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 4 (4) | 7 (9) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 18 (40) | 14 (19) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Condition aggravated (General disorders) | 9 (29) | 29 (65) | 6 (9) | 0 (0)
Fatigue (General disorders) | 0 (0) | 7 (8) | 5 (5) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Local swelling (General disorders) | 3 (8) | 16 (31) | 16 (25) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 12 (17) | 10 (15) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 6 (10) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 6 (9) | 7 (11) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 4 (6) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 3 (7) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 14 (24) | 14 (19) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 4 (5) | 6 (6) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 4 (5) | 5 (10) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (5) | 4 (5) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 3 (4) | 3 (5) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 11 (21) | 11 (13) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (5) | 5 (9) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 7 (15) | 7 (8) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 2 (3) | 17 (41) | 9 (14) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (7) | 6 (10) | 13 (23) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 8 (9) | 5 (7) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (6) | 12 (15) | 5 (9) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 5 (8) | 4 (4) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 8 (10) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 0 (0) | 0 (0) | 11 (15) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 4 (5) | 5 (7) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 6 (22) | 0 (0) | 0 (0)
Urobilinogen urine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (6) | 4 (4) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (5) | 3 (8) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (23) | 25 (69) | 27 (66) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 17 (23) | 8 (12) | 0 (0)
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 6 (6) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (7) | 5 (5) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (13) | 4 (6) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (7) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 15 (20) | 13 (21) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (8) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (10) | 6 (6) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 6 (6) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (15) | 10 (10) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (6) | 8 (8) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (36) | 5 (9) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 9 (10) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (17) | 26 (52) | 23 (46) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 7 (11) | 5 (10) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 15 (28) | 13 (19) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 6 (7) | 5 (8) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 6 (6) | 7 (9) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (3) | 3 (3) | 6 (7) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 5 (8) | 5 (8) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 7 (9) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5) | 4 (4) | 0 (0)
Irritability (Psychiatric disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (6) | 6 (8) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 9 (12) | 6 (8) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 14 (17) | 10 (11) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 4 (8) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 10 (16) | 5 (9) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (14) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (15) | 5 (9) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 3 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (5) | 7 (8) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 26 (30) | 20 (25) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (8) | 6 (7) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (6) | 4 (5) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7) | 3 (8) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (8) | 12 (21) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (51) | 44 (130) | 38 (86) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 5 (11) | 11 (36) | 6 (11) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 5 (7) | 23 (49) | 16 (29) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 4 (6) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (5) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 5 (7) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (15) | 28 (60) | 18 (29) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 (5) | 21 (30) | 9 (12) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 24 (47) | 16 (32) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8) | 5 (5) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 22 (61) | 19 (37) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 6 (8) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6) | 3 (6) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (8) | 4 (7) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
On 04-Dec-2019, participants <14 years were required to interrupt treatment due to partial clinical hold placed on palovarotene clinical development program by the FDA. On 24-Jan-2020, treatment was temporarily halted in participants 14 years and older in palovarotene FOP trials when futility boundary was crossed at an interim analysis in PVO-1A-301 study. After post-hoc analyses, dosing was re-initiated only in participants 14 years and above who were able and willing to re-start treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT02279095/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT02279095/SAP_001.pdf